CLINICAL TRIAL: NCT00387010
Title: A 4-week Open-Label Study to Evaluate the Effect of Treatment With Fentanyl Buccal Tablets on Pain Anxiety Symptoms When Used for the Management of Breakthrough Pain in Opioid-Tolerant Patients With Chronic Pain
Brief Title: Open-Label Study to Evaluate the Effect of Treatment With Fentanyl Buccal Tablets on Pain Anxiety Symptoms When Used for the Management of Breakthrough Pain
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor felt enough information was available for the exploratory assessment of the effect of treatment with FBT on pain anxiety
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25608/3054/BP/US
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-09

CONDITIONS: Pain; Chronic Pain; Breakthrough Pain
MeSH Terms: conditions — Pain; Chronic Pain; Breakthrough Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fentanyl buccal tablets (Experimental): Successful dose strength for each participant was determined during a titration period of no more than 10 days. Participants used the successful dose of 100, 200, 400, 600, or 800 mcg during the four week open-label treatment period.
  Interventions: Drug: Fentanyl Buccal Tablets

INTERVENTIONS:
Drug: Fentanyl Buccal Tablets — Fentanyl buccal tablets (FBT) placed in the buccal cavity above a rear molar until disintegrated, approximately 14-25 minutes.
  Dose titration: Participants self-administered FBT, starting at 100, 200 or 400 mcg (depending on analgesic used pre-study) and titrated to 600 and 800 mcg as needed. For each breakthrough pain (BTP) episode, participants took a dose, and did not take further study drug if adequate pain relief was achieved. If pain was not controlled within 30 minutes, the same dose level was repeated. If pain relief was inadequate 30 minutes after the second dose, usual rescue medication was taken for that BTP episode. Doses were adjusted until pain relief was adequate and side effects were tolerated.
  Open-label: Once the successful dose of FBT was identified (100, 200, 400, 600, or 800 mcg), participants were dispensed a 4-week supply at the successful dose. Participants were not to use FBT for more than 6 BTP episodes or take more than 8 FBT daily.
  Other Names: Fentora; CEP-25608; Fentanyl citrate

SUMMARY:
The primary purpose of the study is to evaluate the impact of treatment with fentanyl buccal tablets on the anxiety symptoms commonly associated with chronic pain in patients with breakthrough pain (BTP). Other purposes are to assess the management of BTP, to evaluate patient functioning, and to determine any influences on the successful dose achieved.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing to provide written informed consent to participate in this study.
* The patient is 18 through 80 years of age.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, using a medically accepted method of birth control (i.e., barrier method with spermicide, steroidal contraceptive [oral, transdermal, implanted, and injected contraceptives must be used in conjunction with the barrier method], or intrauterine device [IUD]) and agree to continued use of this method for the duration of the study.
* The patient has chronic pain of at least 3 months duration associated with any of the following conditions: cancer, diabetic peripheral neuropathy, postherpetic neuralgia, traumatic injury, complex regional pain syndrome, back pain, neck pain, fibromyalgia (patient has met diagnostic criteria), chronic pancreatitis, or osteoarthritis. Other chronic painful conditions may be evaluated for entry upon discussion with and written approval from the Cephalon medical expert.
* The patient is currently using 1 of the following: at least 60 mg of oral morphine/day, or at least 25 mcg of transdermal fentanyl/hour, or at least 30 mg of oxycodone/day, or at least 8 mg of hydromorphone/day, or an equianalgesic dose of another opioid/day as a stable dose of around-the-clock (ATC) therapy for at least 7 days prior to enrollment in the study.
* The patient reports an average pain intensity score, over the prior 24 hours, of 6 or less (0=no pain through 10=worst pain) for the chronic pain.
* The patient experiences, on average, 1 to 4 BTP episodes per day while taking around-the-clock (ATC) opioid therapy, and on average, the duration of each breakthrough pain (BTP) episode is less than 3 hours.
* The patient currently uses opioid therapy for alleviation of BTP episodes occurring at the location of the chronic pain, and achieves at least partial relief.
* The patient must be willing and able to successfully self-administer the study drug, comply with study restrictions, and return to the clinic for scheduled study visits and a follow-up evaluation as specified in this protocol.

Exclusion Criteria:

* The patient has uncontrolled or rapidly escalating pain as determined by the investigator (ie, the ATC therapy may be expected to change between the first and last treatments with study drug), or has pain uncontrolled by therapy that could adversely impact the safety of the patient or that could be compromised by treatment with study drug.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to any ingredient in the study drug.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse.
* The patient has cardiopulmonary disease that, in the opinion of the investigator, would significantly increase the risk of treatment with potent synthetic opioids.
* The patient has medical or psychiatric disease that, in the opinion of the investigator, would compromise collected data.
* The patient's primary painful condition is headache, including migraine.
* The patient is expected to have surgery during the study, and it is anticipated that the surgery will alleviate the patient's pain.
* The patient has had therapy before study drug treatment that, in the opinion of the investigator, could alter pain or response to pain medication.
* The patient is pregnant or lactating.
* The patient has participated in a previous study with fentanyl buccal tablets.
* The patient has participated in a study involving an investigational drug in the previous 30 days.
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (e.g., regional nerve block) that, in the opinion of the investigator, would compromise the patient's safety or compliance with the study protocol, or compromise collected data.
* The patient is involved in active litigation in regard to chronic pain currently being treated.
* The patient has a positive urine drug screen (UDS) for an illicit substance or a medication not legitimately prescribed to the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Birmingham Pain Center, Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Orange County Clinical Trials, Anaheim, California
  - Vertex Clinical Research, Bakersfield, California
  - Lovelace Scientific Resources, Inc., Beverly Hills, California
  - Synergy Clinical Research Center, National City, California
  - Pain Institute of Santa Monica, Santa Monica, California
  - Integrative Pain Manage Centers, Westminster, Colorado
  - Advanced Diagnostic Pain Treatment Center, New Haven, Connecticut
  - Alliance Medical Research Group, Clearwater, Florida
  - Innovative Research of West Florida, Largo, Florida
  - Lovelace Scientific Resources, Inc., Sarasota, Florida
  - Stedman Clinical Trials, Tampa, Florida
  - Dawsonville Family Medicine, Dawsonville, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - Pain and Rehabilitation Clinic of Chicago, Chicago, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Rehabilitation Associates of Indiana, Indianapolis, Indiana
  - Northwest Indiana Center for Clinical Research, PC, Valparaiso, Indiana
  - ICRI, Inc., Overland Park, Kansas
  - Willis-Knighton Pain Management Center, Shreveport, Louisiana
  - Montana Cancer Specialists, Missoula, Montana
  - Lovelace Scientific Resources Center, Henderson, Nevada
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - SUNY - Stonybrook, Stony Brook, New York
  - Pain Consultants of Oregon, Eugene, Oregon
  - Allegheny Pain Management, PC, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Comprehensive Pain Specialists, PLLC, Hendersonville, Tennessee
  - KRK Medical Research, Richardson, Texas
  - BeXar Clinical Trials, LLC, Richardson, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah

REFERENCES:
- [Result] Webster LR, Messina J, Xie F, Nalamachu S. Effect of fentanyl buccal tablet on pain-related anxiety: a 4-week open-label study among opioid-tolerant patients with chronic and breakthrough pain. J Opioid Manag. 2011 Jul-Aug;7(4):297-308. PMID 21957829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 327 patients with chronic pain and breakthrough pain (BTP) were screened for enrollment into this study. Of the 327 patients screened, 218 patients at 31 centers in the US met entry criteria and were considered eligible for enrollment into the study.
Period: Dose Titration Period
Arm/Group | Fentanyl Buccal Tablets
Started | 218
Completed | 180
Not Completed | 38
Not completed — Adverse Event | 12
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 2
Not completed — Noncompliance with study medication | 8
Not completed — Noncompliance with study procedures | 7
Period: Treatment Period
Arm/Group | Fentanyl Buccal Tablets
Started | 180
Full Analysis Set | 175 (FAS: treated patients with at least 1 paired baseline and post baseline efficacy assessment)
Completed | 169
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1
Not completed — Noncompliance with study medication | 2
Not completed — Noncompliance with study procedures | 3
Not completed — Participant reported study drug stolen | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 218
Age Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124
  Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 203
  Unknown or Not Reported | 11
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 208
  Unknown or Not Reported | 1
Primary chronic painful condition [Number; unit: participants]
  Back pain | 136
  Neck pain | 14
  Fibromyalgia | 13
  Traumatic injury | 12
  Osteoarthritis | 11
  Complex regional pain syndrome | 9
  Diabetic peripheral neuropathy | 3
  Cancer | 3
  Chronic pancreatitis | 2
  Other | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Pain Anxiety Symptoms Scale (PASS) Total Score at Approximately Week 5
Description: The change from baseline to approximately week 5 in the PASS total score. PASS asks participants to indicate how often they engage in each of the 40 thoughts or activities that represent anxiety symptoms on a scale of 0=never to 5=always. The total score has a range of 0-200.
Time Frame: Day 0 (baseline), approximately week 5
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
units on a scale | -1.6 (20.71)
Statistical Analysis 1: Comparison: Fentanyl Buccal Tablets; Test type: Superiority or Other; p = 0.3223, t-test, 2 sided; Mean Difference (Net) = -1.6, 95% CI 2-sided [-4.64 to 1.54]

2. Secondary Outcome: Change From Baseline in the Pain Anxiety Symptoms Scale (PASS) Subscale Scores at Approximately Week 5
Description: The change from baseline to approximately week 5 in the PASS subscale scores. PASS asks participants to indicate how often they engage in each of the 40 thoughts or activities that represent anxiety symptoms on a scale of 0=never to 5=always. Those 40 questions are organized into four subscales: fear, cognitive anxiety, somatic anxiety, and escape/avoidance. Each subscale score is obtained by summing the answers to the ten items in the subscore resulting in a range of 0-50.
Time Frame: Day 0 (baseline), approximately week 5
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
units on a scale
  Fear | -0.5 (6.14)
  Cognitive anxiety | -1.1 (7.20)
  Somatic anxiety | 0.4 (7.39)
  Escape/avoidance | -0.4 (5.87)

3. Secondary Outcome: Change From Baseline in the Beck Depression Inventory at Approximately Week 5
Description: Change from baseline to endpoint (week 4 of Treatment period or last post baseline visit) in the Beck Depression Inventory (BDI). The BDI is a self-reporting instrument that asks 21 questions regarding how the participant felt in the past few days. Answers are in sentence form, and offer a scale where the first answer (worth 0 points) indicates no depression and the fourth answer (worth 3 points) indicates significant depression. Totals (0-63) are grouped so that totals of 1-10 are interpreted as 'These ups and downs are considered normal' and scores >40 indicate extreme depression.
Time Frame: Day 0 (baseline), approximately week 5
Population: Full analysis set of participants who answered the questions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 169
units on a scale | -1.1 (6.98)

4. Secondary Outcome: Change From Baseline in the West Haven-Yale Multidimensional Pain Inventory Subscales at Approximately Week 5
Description: Change from baseline to endpoint (week 4 of Treatment period or last post baseline visit) in the Multidimensional Pain Inventory Subscales. Answers to questions in the MPI are captured on a 7-point scale, with 0=most positive answer and 6= least positive answer. Twenty questions focus on pain, fourteen on a significant other's response when participant is in pain, and eighteen questions about daily activities. There are a total of 13 subscales with variable ranges. Subscales and corresponding ranges are listed in the results table. The General Activity category combines the Household Chores, Outdoor Work, Activities Away from Home, and Social Activities categories.
Time Frame: Day 0 (baseline), approximately week 5
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
units on a scale
  Interference (0-54) | -0.2 (0.90)
  Support (0-18) | -0.0 (1.02)
  Pain Severity (0-18) | -0.3 (0.97)
  Life-Control (0-12) | 0.1 (1.25)
  Affective Distress (0-18) | -0.1 (1.24)
  Negative Responses (0-24) | -0.1 (1.01)
  Solicitous Responses (0-24) | 0.1 (1.03)
  Distracting Responses (0-36) | 0.2 (1.02)
  Household Chores (0-30) | 0.1 (1.05)
  Outdoor Work (0-30) | -0.0 (0.74)
  Activities Away from Home (0-24) | 0.1 (0.87)
  Social Activities (0-24) | 0.0 (0.86)
  General Activity (0-108) | 0.0 (0.67)

5. Secondary Outcome: Medication Preference From the Pain Flare Treatment Satisfaction Questionnaire at Approximately Week 5
Description: The summary question from the Pain Flare Treatment Satisfaction Questionnaire asked participants which medication they preferred to use for their break-through pain. Options were 1) Prior medication 2) Study medication 3) no preference
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the questions.
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 174
participants
  Prior medication | 38
  Study medication | 115
  No preference | 21

6. Secondary Outcome: Patient Assessment of Ability to Go to Work at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) participants completed the Patient Assessment of Function Scale which asks 7 questions about the effect of study treatment on the patient's ability to function. This question asks about the ability to go to work.
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the question
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 88
participants
  Very much worsened | 2
  Much worsened | 0
  Slightly worsened | 2
  Unchanged | 51
  Slightly improved | 14
  Much improved | 13
  Very much improved | 6

7. Secondary Outcome: Patient Assessment of Ability to Perform at Work at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) participants completed the Patient Assessment of Function Scale which asks 7 questions about the effect of study treatment on the patient's ability to function. This question asks about the ability to perform at work and includes both work outside the home and housework.
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the question
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 4
  Much worsened | 1
  Slightly worsened | 6
  Unchanged | 69
  Slightly improved | 41
  Much improved | 45
  Very much improved | 9

8. Secondary Outcome: Patient Assessment of Ability to Walk at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) participants completed the Patient Assessment of Function Scale which asks 7 questions about the effect of study treatment on the patient's ability to function. This question asks about the ability to walk.
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the question
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 174
participants
  Very much worsened | 3
  Much worsened | 1
  Slightly worsened | 5
  Unchanged | 76
  Slightly improved | 42
  Much improved | 36
  Very much improved | 11

9. Secondary Outcome: Patient Assessment of Ability to Exercise at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) participants completed the Patient Assessment of Function Scale which asks 7 questions about the effect of study treatment on the patient's ability to function. This question asks about the ability to exercise.
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the question
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 3
  Much worsened | 1
  Slightly worsened | 5
  Unchanged | 90
  Slightly improved | 46
  Much improved | 21
  Very much improved | 9

10. Secondary Outcome: Patient Assessment of Ability to Participate in Social Events at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) participants completed the Patient Assessment of Function Scale which asks 7 questions about the effect of study treatment on the patient's ability to function. This question asks about the ability to participate in social events.
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the question
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 1
  Much worsened | 3
  Slightly worsened | 6
  Unchanged | 80
  Slightly improved | 46
  Much improved | 34
  Very much improved | 5

11. Secondary Outcome: Patient Assessment of Ability to Have Sex at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) participants completed the Patient Assessment of Function Scale which asks 7 questions about the effect of study treatment on the patient's ability to function. This question asks about the ability to have sex.
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the question
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 173
participants
  Very much worsened | 4
  Much worsened | 2
  Slightly worsened | 3
  Unchanged | 129
  Slightly improved | 18
  Much improved | 12
  Very much improved | 5

12. Secondary Outcome: Patient Assessment of Ability to Enjoy Life at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) participants completed the Patient Assessment of Function Scale which asks 7 questions about the effect of study treatment on the patient's ability to function. This question asks about the ability to enjoy life.
Time Frame: approximately week 5
Population: Full analysis set of participants who answered the question
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 2
  Much worsened | 1
  Slightly worsened | 6
  Unchanged | 66
  Slightly improved | 48
  Much improved | 38
  Very much improved | 14

13. Secondary Outcome: Clinical Assessment of Patient Function - General Activities - at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) investigators completed the Clinical Assessment of Patient Function Scale which asks 5 questions about the effect of study treatment on the patient's ability to function. This question asks about the patient's general activities.
Time Frame: approximately week 5
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 0
  Much worsened | 1
  Slightly worsened | 4
  Unchanged | 58
  Slightly improved | 57
  Much improved | 46
  Very much improved | 9

14. Secondary Outcome: Clinical Assessment of Patient Function - Patient's Walking Ability - at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) investigators completed the Clinical Assessment of Patient Function Scale which asks 5 questions about the effect of study treatment on the patient's ability to function. This question asks about the patient's walking ability.
Time Frame: approximately week 5
Population: Full analysis set. One participant was not assessed by the investigator.
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 174
participants
  Very much worsened | 0
  Much worsened | 0
  Slightly worsened | 4
  Unchanged | 81
  Slightly improved | 48
  Much improved | 31
  Very much improved | 10

15. Secondary Outcome: Clinical Assessment of Patient Function - Patient's Ability to Work/Perform Activities of Daily Living - at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) investigators completed the Clinical Assessment of Patient Function Scale which asks 5 questions about the effect of study treatment on the patient's ability to function. This question asks about the patient's ability to work and perform activities of daily living.
Time Frame: approximately week 5
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 0
  Much worsened | 1
  Slightly worsened | 5
  Unchanged | 63
  Slightly improved | 55
  Much improved | 39
  Very much improved | 12

16. Secondary Outcome: Clinical Assessment of Patient Function - Patient's Relationship With Others - at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) investigators completed the Clinical Assessment of Patient Function Scale which asks 5 questions about the effect of study treatment on the patient's ability to function. This question asks about the patient's relationship with others.
Time Frame: approximately week 5
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 0
  Much worsened | 0
  Slightly worsened | 1
  Unchanged | 98
  Slightly improved | 35
  Much improved | 32
  Very much improved | 9

17. Secondary Outcome: Clinical Assessment of Patient Function - Patient's Enjoyment of Life - at Approximately Week 5
Description: At the endpoint of the study (week 4 of Treatment period or last post baseline visit) investigators completed the Clinical Assessment of Patient Function Scale which asks 5 questions about the effect of study treatment on the patient's ability to function. This question asks about the patient's enjoyment of life.
Time Frame: approximately week 5
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 175
participants
  Very much worsened | 0
  Much worsened | 2
  Slightly worsened | 1
  Unchanged | 69
  Slightly improved | 45
  Much improved | 43
  Very much improved | 15

18. Secondary Outcome: Summary of Participants' Successful Dosing Levels of Fentanyl Buccal Tablets to Control Episodes of Breakthrough Pain (BTP)
Description: During the dose titration period, participants self-administered FBT, starting at 100, 200 or 400 mcg (depending on analgesic used pre-study) and titrated to 600 and 800 mcg if needed. For each breakthrough pain (BTP) episode, participants took a dose, and did not take further study drug if adequate pain relief was achieved. If pain was not controlled within 30 minutes, the same dose level was repeated. If pain relief was inadequate 30 minutes after the second dose, usual rescue medication was taken for that BTP episode. Doses were adjusted until pain relief was adequate and side effects were tolerated. This outcome summarizes the successful dose levels identified during the titration period.
Time Frame: up to 10 days
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Fentanyl Buccal Tablets
Number analyzed (Participants) | 218
participants
  100 mcg | 18
  200 mcg | 49
  400 mcg | 41
  600 mcg | 31
  800 mcg | 41
  None (no successful dose) | 38

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events: Day 1 to approximately 5 weeks.
Arm/Group | Fentanyl Buccal Tablets
Serious Adverse Events (participants affected / at risk) | 4/218
Other Adverse Events (participants affected / at risk) | 21/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Buccal Tablets (N=218)
Bronchitis (Infections and infestations) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Buccal Tablets (N=218)
Nausea (Gastrointestinal disorders) | 21

LIMITATIONS AND CAVEATS:
This study was terminated early. Additional research is recommended to develop a valid measure of anxiety, specifically related to breakthrough pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.